CLINICAL TRIAL: NCT06248918
Title: The Effects of a Nurse-led Using Wearable Technology Physical Activity Program on Health-Related Quality of Life and Physical Activity Level Among Breast Cancer Survivors
Brief Title: Nurse-led Physical Activity Program Among Breast Cancer Survivors
Acronym: WATSOCPAP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, sura kaya, Research Assistant, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IMUH-HEM-SK-01
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer Female; Survivorship; Health Behavior
Keywords: Breast Cancer; Survivors; Physical Activity; Social Cognitive Theory; Health-Related Quality Of Life
MeSH Terms: conditions — Health Behavior; Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will receive an exercise plan, activity tracker, and physical activity coaching program based Social Cognitive Theory.
  Interventions: Behavioral: WATSOCPAP
- Control Group (No Intervention): The control group will not take any intervention but take a standard care, the post-tests will be collected at the end of 12 weeks.

INTERVENTIONS:
Behavioral: WATSOCPAP — Participants will receive an supervised and individualized exercise plan, activity tracker, and physical activity coaching program based Social Cognitive Theory. Participants will be administered strengthening and aerobic exercise program, structured and individualized according to the person's individual capacity and needs, under the supervision of a physiotherapist. The activity tracker will provide real-time activity information about daily steps, time spent with MVPA (minutes/day) and sedentary time. The nurse-led physical activity coaching program was planned according to the Social Cognitive Theory (SCT) components such as self-regulation, outcome expectation, social support and perceived environment. The interventions will continue with online and the 12-week program will be completed.
  Arms: Intervention Group

SUMMARY:
A nurse-led physical activity program including an individualized exercise program using wearable technology and health coaching based on Social Cognitive Theory will be implemented for women surviving cancer. The impact of the nurse-led physical activity program on physical activity level, health-related quality of life and cognitive factors (self regulation, outcome expectation, self efficacy, perceived social support, perceived environment) will be evaluated in the study.

DETAILED DESCRIPTION:
This study protocol describes a randomized controlled trial with parallel group design. Participants will be Breast cancer survivors who aged 18-65, have finished active treatment (surgery, chemotherapy, and/or radiotherapy) in the previous 5 years, no evidence of recurrence and contraindications, and are completing less than 150-minutes of Moderate-Vigorous intensity Physical Activity (MVPA) per week. Participants will be randomly assigned to the intervention and control group.

Wearable Technology using Social Cognitive Theory based physical activity program (WATSOCPAP) created for the Intervention Group includes 3 different intervention components: (1) Supervised and individualized exercise plan; (2) Physical activity monitoring with activity tracker; (3) Nurse-led physical activity coaching program. Participants will be administered strengthening and aerobic exercise program, structured and individualized according to the person's individual capacity and needs, under the supervision of a physiotherapist. The activity tracker will provide real-time activity information about daily steps, time spent with MVPA (minutes/day) and sedentary time. The nurse-led physical activity coaching program was planned according to the Social Cognitive Theory (SCT) components such as self-regulation, outcome expectation, social support and perceived environment. WATSOCPAP is a 12-week program that includes text messages, face-to-face and online interviews. The first intervention in this group will begin with a 60-minute face-to-face individual training. After the first interview, text messages will be made according to the Social Cognitive Theory (SCT) components per weeks. Control group will receive standard care. Follow-up questionnaires will be applied by repeating the post-test at the 24th week. In the intervention and control groups, post-test will be applied 12 weeks after the pre-test, and follow-up questionnaires will be applied 24 weeks after the pre-test.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65
* Female gender
* Diagnosed with stage I-III breast cancer survivors,
* Completed active cancer primary treatment (surgery, chemotherapy, and/or radiotherapy) in the previous 5 years, excluding hormone therapy,
* No evidence of recurrence,
* No contraindications,
* Less than 150 minutes of moderate-intensity physical activity or 75 minutes of vigorous-intensity physical activity per week,
* Having a smart mobile phone and to access and use the internet,
* Live in Istanbul city,
* No medical condition(s) that non-adherence to an exercise program

Exclusion Criteria:

* Currently pregnant or planning to become pregnant during the study period,
* Musculoskeletal, neurological, respiratory, metabolic or cardiovascular health problems which preclude exercise,
* Cancer recurrence and resumption of active cancer treatment.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Self Reported Physical Activity | Baseline, 12 weeks, 24 weeks
  Change in physical activity, as measured by the "International Physical Activity Questionnaire-Short Form", from baseline to 12 and 24 weeks. Participants report frequency of light, moderate and vigorous physical activity, and average duration (minutes/week) bouts for 10 minutes or longer in the last seven days. Scores for light, moderate and vigorous exercise are combined to compute total physical activity minutes/week. Computation of the total score for the short form requires summation of the duration (in minutes) and frequency (days) of walking, moderate-intensity and vigorous-intensity activities. Standard MET (metabolic equivalent) values for activities were established. The 'MET-min/week' value is obtained by multiplying the MET value of each physical activity level with the days and minutes this physical activity is performed every week. The obtained MET value is classified as HEPA active (MET>3000), minimally active (MET=600-3000), and inactive (MET<600).

SECONDARY OUTCOMES:
Health Related Quality of Life: EORTC-QLQ-C30 | Baseline, 12 weeks, 24 weeks
  Change in general health-related quality of life, as measured using the The European Organization for Research and Treatment of Cancer (EORTC) developed a cancer-specific core questionnaire (QLQ-C30), from baseline to 12 and 24 weeks. QLQ-C30 is composed of 30 items assessing global perceived health status and QoL. These items are grouped in five functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning); three symptom scales (fatigue, nausea & vomiting, and pain); six single item scales. Responses are coded on a scale of 0 to 4 where 0 is not at all and 4 is very much. A rise in the functional dimension score and a fall in the symptom dimension score signify an improvement in QoL. High general well-being dimension scores are indicative of a QoL. The computation yields scores for every dimension out of a possible 100, with scores ranging from 0 to 100.
Health Related Quality of Life-Breast Cancer Specified: EORTC-QLQ-BR23 | Baseline, 12 weeks, 24 weeks
  Change in health-related quality of life-Breast Cancer Specified, as measured using the EORTC-QLQ-BR23, from baseline to 12 and 24 weeks. QLQ-BR23 questionnaire has 23 items to assess functional scales (body image), sexual functioning, sexual enjoyment, and future perspective); symptom scales (systemic therapy side effects, breast symptoms, arm symptoms, and upset by hair loss). The total score range of the scale is 0-100. A high quality of life is indicated by a low score in the symptom dimension and a high score in the functional dimension of the scale.
BMI | Baseline, 12 weeks, 24 weeks
  Change in BMI, as measured objectively with digital scales, from baseline to to 12 and 24 weeks.
Fatigue | Baseline, 12 weeks, 24 weeks
  Change in fatigue, as measured by the The Functional Assessment of Chronic Illness Treatment-Fatigue Scale (FACIT-F), from baseline to 12 and 24 weeks. The FACIT-F Scale is composed of 13 expressions that measure the fatigue that the patients had in the last seven days.7 The expressions on the scale consist of Likert type question form which is scored between 0 and 4 and con- sists of ''Not at all'', ''A little bit'', ''Somewhat'', ''Quite a bit'', and ''Very much''. The total score range of the scale is 0-52. The higher the scale score, the lower the fatigue level of the patient.
Self-efficacy For Exercise | Baseline, 12 weeks, 24 weeks
  Change in self-efficacy for exercise, as measured by the The Exercise Self-efficacy Scale, from baseline to 12 and 24 weeks. Responses 18 items, ranging from 0 (cannot do it) to 100 (definitely can do it), are summed, with higher values representing higher efficacy beliefs for exercises.
Outcome Expectations for Exercise | Baseline, 12 weeks, 24 weeks
  Change in outcome expectations for exercise, as measured by the Multidimensional Outcome Expectations for Exercise Scale, from baseline to 12 and 24 weeks. Responses for three subscales (physical subscale, social subscale, self-evaluative subscale), ranging from 1 (strongly disagree) to 5 (strongly agree), are summed, with higher values representing higher outcome expectations for exercise.
Self-regulation | Baseline, 12 weeks, 24 weeks
  Change in self-regulation, as measured using by self-report questionnaire, from baseline to 12 and 24 weeks. Responses to two subscales (Exercise goal-setting, Exercise planning and scheduling), ranging from 1 (does not describe) to 5 (describes completely), are averaged to yield two subscales. Higher subscale scores represent higher self-regulation.
Multidimensional Perceived Social Support Scale | Baseline, 12 weeks, 24 weeks
  Change in social support, as measured by the Multidimensional Perceived Social Support Scale, from baseline to 12 and 24 weeks. Responses for three factors (Family participation, Friend participation, a special person participation), ranging from 1 to 7, are summed, with higher values representing higher perceived social support.
Perceived Environment | Baseline, 12 weeks, 24 weeks
  Change in perceived environment, as measured using the Physical Activity Neighborhood Environment Scale (PANES) survey, from baseline to 12 and 24 weeks. PANES is a 17-item measure perceived attributes of the neighborhood environment related to physical activity. Concepts assessed by PANES include residential density (1 item), access to destinations (3 items), pedestrian and bicycling facilities (4 items), recreational facilities (1 item), aesthetic qualities (1 item), social environment (1 item), street connectivity (1 item), traffic safety (2 items), crime safety (2 items), and household motor vehicles (1 item). With the exception of the residential density and household motor vehicle questions, items ranging ranging from 1 (strongly disagree) to 5 (strongly agree), as well as don't know or doesn't apply response option.

CONTACTS AND LOCATIONS:
Overall Officials: Sura Kaya, MSc, Principal Investigator — Medipol University
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol was planned to share in one year with other researchers.
Supporting Information: Study Protocol
Time Frame: One year
Access Criteria: Individual participants data that underlie the results reported in this article, after de identification (text, tables, figures, appendices).